CLINICAL TRIAL: NCT03931603
Title: Endometriosis of the Recto-sigmoid: MRI Criteria Predictive of Shaving or Segmental Resection
Brief Title: Endometriosis of the Recto-sigmoid: MRI (Magnetic Resonance Imaging) Criteria Predictive of Shaving or Segmental Resection
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 17-170
Record Dates: First submitted 2018-11-15; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Endometriotic Parietal Involvement of the Rectosigmoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI — MRI protocol associating sagittal and axial (+/- coronal) sequences in T2 + / - turbo spin T1 weighting with fat saturation.

SUMMARY:
Evaluate MRI criteria predictive of the type of surgery to be performed for an "in sano" resection of endometriotic involvement of the recto-sigmoid by a resection without opening of the rectal mucosa ("shaving") versus a segmental resection.

DETAILED DESCRIPTION:
PURPOSE: To retrospectively determine the accuracy of MRI rectal and pararectal signs in predicting a segmental resection of lesions located in the rectum until the recto-sigmoid junction.

MATERIALS AND METHODS: Institutional review board approval for this study was obtained and waived written informed consent. The MR images of 61 patients treated for rectal endometriosis over a 6 years period were reviewed. Two blinded readers performed in consensus a systematic analysis of 7 rectal (length, transverse axis, thickness and circumference of the lesion, and presence of a convex base, submucosal edema and hyperintense cystic areas) and 4 pararectal (posterior vaginal fornix, parametrial, ureteral and sacro-recto-genital septum involvements) signs for each lesion. MR imaging results were compared with surgical procedure (shaving versus segmental resection). Efficacy parameters were calculated with 95 % confidence intervals (CIs).

ELIGIBILITY:
Inclusion Criteria:

* operated patient for a pelvic endometriosis with resection without opening of the rectal mucosa ("shaving") or with segmental resection of the recto-sigmoidienne.
* Performing a preoperative pelvic MRI with at least 2 perpendicular T2 planes

Exclusion Criteria:

* Refusal to use clinical data and exploration acquired
* Absence of interpretable preoperative pelvic MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients treated in the gynecological surgery departments of the University Hospital Center of the Civil Hospitals of Lyon: Lyon Sud.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Comparison of MRI data with intraoperative data and anatomopathology | Intraoperatively
  MRI criteria of parietal involvement will be confronted with the type of surgery performed (shaving or segmental resection) A rectosigmoid parietal involvement will be defined by the nodular replacement of the normal signal of the digestive muscularis, on at least two planes of cuts or two different weightings.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Centre Hospitalier Lyon Sud -Service de Radiologie, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No